CLINICAL TRIAL: NCT00312741
Title: Prospective Study on Benefits Derived From Microbiological Tests in Community-Acquired Pneumonia
Brief Title: Usefulness of Microbiological Tests in Community-Acquired Pneumonia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Arnau de Vilanova (Other)
Other Study IDs: pneumonia1
Record Dates: First submitted 2006-04-07; First posted 2006-04-11 (Estimated); Last update posted 2009-02-27 (Estimated); Status verified 2009-02

CONDITIONS: Community-Acquired Pneumonia
Keywords: community-acquired pneumonia; microbiological tests; urinary antigen; selection of antibiotic treatment
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: empirical versus microbiological guided treatment

SUMMARY:
The hypothesis is that community-acquired pneumonia is usually a monomicrobial infection. Therefore, early detection of the etiology allows to select the most active, narrow-spectrum, and cheap, and less toxic antibiotic agent.

DETAILED DESCRIPTION:
In community-acquired pneumonia, identification of the etiologic agent has theoretically important advantages. For individual patients, it facilitates the administration of a targeted, narrow-spectrum antibiotic therapy that may improve the efficacy of treatment, and reduces risks of antibiotic-related toxicity. For the community, microbiologic results contribute to understanding the local microbial epidemiology of community-acquired pneumonia and the antimicrobial resistance patterns of pathogens, information that is essential in the instauration or modification of empiric treatment regimens.

Guidelines recommend that all admitted patients with community-acquired pneumonia should have a collection of two sets of blood cultures, a good quality sputum sample for Gram stain and culture, a sample of pleural fuid if present and, for severe patients, an urine sample for antigen detection. In contrast, several prospective studies (usually without include urinary tests) concluded that these microbiological studies have limited value in the management of patients admitted with community-acquired pneumonia.

In addition, microbiological studies could provide erroneous or incomplete information. Thus, investigations has showed false-positive results from pneumococcal antigen detection in urine caused by a frequent persistence of positivity after infection or a nasopharyngeal or bronchial colonization. Other authors suggested that community-acquired pneumonia is a polymicrobial infection; consequently, despite the detection of a true microorganism, treatment needs to be also addressed against other potential pathogenic agents.

The purpose of the study is to assess the clinical and the economic derived from the initial microbiological studies, including antigen detection tests in urine for Streptococcus pneumoniae and Legionella pneumophila, in patients with community-acquired pneumonia.

The hypothesis is that community-acquired pneumonia is usually a monomicrobial infection. Therefore, early detection of the etiology allows to select the most active, narrow-spectrum, and cheap, and less toxic antibiotic agent.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years and above
* Clinical and radiological diagnosis of community-acquired pneumonia
* Informed consent of patient
* Hospital admission

Exclusion Criteria:

* Prior hospital admission (less than 15 days)
* Alternative diagnosis at the discharge
* Immunosuppression (HIV infection, immunosuppressive therapies, neutropenia)
* Risk factors for unusual etiologies
* Patient is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2006-04; Study Completion 2008-05 (Estimated)

PRIMARY OUTCOMES:
Clinical and economic consequences obtained with the antibiotic selection in basis to early mcrobiological results

SECONDARY OUTCOMES:
Importance of polimicrobial etiology in community-acquired pneumonia
Practice usefulness of urinary antigen detection tests in pneumonia

CONTACTS AND LOCATIONS:
Overall Officials: Miquel Falguera, M.D., Principal Investigator — Hospital Arnau de Vilanova (Lleida)
Locations (1):
- Hospital Arnau de Vilanova, Lleida, Lleida, Spain